CLINICAL TRIAL: NCT02967601
Title: Influence of Preoperative Anxiety on Shivering During Elective Caesarean Section Under Spinal Anaesthesia
Status: Completed | Type: Observational
Sponsor: Bartłomiej Wódarski (Other)
Responsible Party: Sponsor-Investigator, Bartłomiej Wódarski, MD, Centre of Postgraduate Medical Education
Organization: Centre of Postgraduate Medical Education (Other)
Other Study IDs: shiv01
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Shivering
Keywords: shivering, cesarean section, anxiety, STAI
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective Cesarean Section
  Interventions: Behavioral: STAI (State Trait Anxiety Inventory) questionaire

INTERVENTIONS:
Behavioral: STAI (State Trait Anxiety Inventory) questionaire — Each patient would fill the STAI questionaire before Cesarean Section (on the same day, in the morning)

SUMMARY:
Background Shivering occurs in circa 50 percent of cases during caesarean section under spinal anesthesia. The phenomenon's reasons and its mechanism are unclear, and while it does not endanger the patients' health, the sensations proved to be unpleasant and a subject of a number of patients' complains.

Objectives The main objective of the study is to establish the anxiety factors that influence the risk of muscle-shivering and a detailed assessment of the probability of existence of the link between increased anxiety levels with the shivering in case of patients undergoing the elective caesarean section.

Moreover, the outcomes of the study could help to further understand the phenomenon, reduce its occurence and as a result of that - improve the comfort of the patients in the perioperative period, as well as reduce the frequency of pharmacological treatment to halt the symptoms of muscle shivering.

Methodology Patients would be asked to fill the STAI (State - Trait Anxiety Inventory) questionaire in the morning preceding the surgery. Results would be interpreted by one of the investigators, who obtained a masters degree in psychology. Caesarean section under spinal anesthesia would be performed according to standard procedures used in the Samodzielny Publiczny Szpital Kliniczny Centrum Medyczne Kształcenia Podyplomowego (SPSK CMKP) hospital, with standard non-invasive monitoring (HR, noninvasive blood pressure (NIBP), oxygen saturation (SpO2), Temperature). Additionally, the anesthesiologist would note the incidence of shivering and its precise timing 1. since the spinal block 2. since the child-birth. Moreover, patients would rate anesthesiology team influence on her anxiety level during the cesarean section in 5 grade scale - data would be collected by psychologist.

The survey is planned for a one year timespan or until 200 patients have enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 y.o.
* ASA 1-2
* signed informed consent form after reading the information about the study and talking with one of the investigators

Exclusion Criteria:

* conversion to general anesthesia
* any severe obstetric complications, which affects obstetric or anesthesiology procedure
* severe bleeding
* language barrier
* anxiolytic/psychotropic drugs use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing an Elective Ceasearean Section, qualified for spinal anaesthesia with American Society of Anesthesiologists (ASA) physical status classification system I-II.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Correlation between shivering and anxiety (STAI score) | during elective cesarean section

SECONDARY OUTCOMES:
Correlation between shivering and patient's temperature (noninvasive) | during elective cesarean section
Correlation between shivering and patient's subjective assesment of anesthesiology team attitude | during elective cesarean section
Correlation between shivering and patient's obstetric history socio-economical data. | during elective cesarean section

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny im. prof. W. Orłowskiego w Warszawie, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No